CLINICAL TRIAL: NCT03125252
Title: Impact of Non-pharmacological Prevention Measures on the Incidence of Delirium in Adult Intensive Care Units
Acronym: DELIREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15 7842 16
Record Dates: First submitted 2017-03-05; First posted 2017-04-24 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Delirium
Keywords: Delirium; Reanimation; Conversational hypnosis
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bundle (Experimental): Specific action plan : ABCDE, complemented with care related to the nursing and paramedical role concerning the patient's environmental factors
  Interventions: Other: Bundle
- Control (Other): Standard paramedical and medical practices
  Interventions: Other: Standard Paramedical and Medical practices

INTERVENTIONS:
Other: Bundle — Awakening and Breathing Coordination Delirium monitoring and management (detection and management of delirium) Early mobility
  Factors of environment:
  * thirst
  * noise
  * pain and well-being
  * sleep
  * isolation
  Other Names: ABCDE
  Arms: Bundle
Other: Standard Paramedical and Medical practices — The current recommendations recommend the following scheme:
  * Identification and correction of an organic cause / factors (sepsis, metabolic disorders, withdrawal syndrome, pain)
  * Use of non-pharmacological means (early mobilization, correction of sensory deficits, temporo-spatial reorientation strategies)
  * Use of reference antipsychotic pharmacological means
  Arms: Control

SUMMARY:
The main objective is to evaluate the impact of the "bundle of actions" on the delirium's incidence in resuscitation patients during their stay in the service, compared to a conventional treatment.

The investigators therefore hypothesize that a set of coordinated paramedical actions in the prevention of delirium would reduce its incidence by 15% compared to conventional care.

DETAILED DESCRIPTION:
The "Bundle of Actions" is a coordinated and specific action plan, which has already been validated, focusing on the coordination of wake-up and respiration, the management of delirium, as well as the early mobility of the patient. Innovation consists of simple, reproducible nursing care that reduces triggers of delirium; as well as the use of two new approaches in reanimation: conversational hypnosis and early and comprehensive re-empowerment of the patient in the management of his pain and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the trusted person and the patient upon waking
* Hospitalized in reanimation service (first hospitalization or transfer of another service)
* 48 hours of sedation with intubation during hospitalization (all combinations of morphine, hypnotics, sedatives, anesthetics, narcoleptics)
* Francophone (able to understand all evaluations)

Criteria for the inclusion of 50 delirium positive patients drawn from the Toulouse center (participating in the neuropsychological evaluation): In addition to those mentioned above:

* Absence of pre-existing cognitive impairment (patients whose relative has completed the IQCode questionnaire and whose score is <3.4 points)
* Visual, auditory (authorized equipment) skills and adequate oral or written expression for the proper conduct of neuropsychological tests.

Exclusion Criteria:

* Pregnant women
* Evolutive neurological disease leading to cognitive impairment (multiple sclerosis, Parkinson's disease, Alzheimer's disease), and / or focal neurological disease leading to cognitive impairment (head trauma, stroke, ...)
* Evolving psychiatric illness (including severe depression)
* Voluntary drug poisoning
* Patients who have already participated in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Incidence rate of delirium | Day 60
  CAM-ICU Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) scale.

SECONDARY OUTCOMES:
Duration of the delirium between the diagnosis and the resolution of the delirium | Day 60
  The duration of the delirium (in days) between the diagnosis and the resolution of the delirium will be done until 60 days of the stay of the patients in intensive care.
Evaluation of cognitive and psycho-behavioral functions. | Day 60 and month 3
  Cognitive and psycho-behavioral functions are usually evaluated by a corpus of test :
  * memory : Test of 5 words and Free Recall Test
  * executive : Fast Evaluation Battery for Executive Functions, Trail Making Test, Digit Span, Stroop and Verbal Fluences and Animals
  * praxis : Mahieux's Test
  * language : D0 80
  * behavior : Montgomery's scale (depression), Starkstein's scale (apathy).
Quality of life at one year | Year 1
  The evaluation of 142 first patients delirium positive: the first 12 patients delirium positive in the 6 centers of the arm to which Toulouse will not belong, and the first 14 patients delirium positive in the 5 centers of the arm to which Toulouse will belong (Toulouse excluded), 1 year after the date of their inclusion in the study during their hospitalization in reanimation service.
  This evaluation of Quality of life of the first patients detected positive to delirium will be carried out using the validated French standardized questionnaire or Short Form 36 item (SF-36) which will be sent by post to the patient's home.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny CROZES, nurse, Study Director — University Hospital, Toulouse
Locations (14):
- France (14):
  - Saint-André Hospital, Bordeaux
  - Hospital Castres-Mazamet, Castres
  - Estaing Hospital, Clermont-Ferrand
  - Gabriel Montpied, Clermont-Ferrand
  - Nord Hospital, Marseille
  - Saint-Joseph Hospital, Marseille
  - Montauban Hospital, Montauban
  - Hospital, Montpellier
  - Caremeau Hospital, Nîmes
  - Perpignan Hospital, Perpignan
  - Jacques Puel Hospital, Rodez
  - University Hospital Toulouse, Toulouse
  - Oncologic Hospital, Toulouse
  - Rangueil Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aissaoui Y, Zeggwagh AA, Zekraoui A, Abidi K, Abouqal R. Validation of a behavioral pain scale in critically ill, sedated, and mechanically ventilated patients. Anesth Analg. 2005 Nov;101(5):1470-1476. doi: 10.1213/01.ANE.0000182331.68722.FF. PMID 16244013
- [Background] Arend E, Christensen M. Delirium in the intensive care unit: a review. Nurs Crit Care. 2009 May-Jun;14(3):145-54. doi: 10.1111/j.1478-5153.2008.00324.x. PMID 19366412
- [Background] Balas MC, Vasilevskis EE, Burke WJ, Boehm L, Pun BT, Olsen KM, Peitz GJ, Ely EW. Critical care nurses' role in implementing the "ABCDE bundle" into practice. Crit Care Nurse. 2012 Apr;32(2):35-8, 40-7; quiz 48. doi: 10.4037/ccn2012229. PMID 22467611
- [Background] Chanques G, Payen JF, Mercier G, de Lattre S, Viel E, Jung B, Cisse M, Lefrant JY, Jaber S. Assessing pain in non-intubated critically ill patients unable to self report: an adaptation of the Behavioral Pain Scale. Intensive Care Med. 2009 Dec;35(12):2060-7. doi: 10.1007/s00134-009-1590-5. PMID 19697008
- [Background] Devlin JW, Brummel NE, Al-Qadheeb NS. Optimising the recognition of delirium in the intensive care unit. Best Pract Res Clin Anaesthesiol. 2012 Sep;26(3):385-93. doi: 10.1016/j.bpa.2012.08.002. PMID 23040288
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Erickson MH, Rossi EL. Two level communication and the microdynamics of trance and suggestion. Am J Clin Hypn. 1976 Jan;18(3):153-71. doi: 10.1080/00029157.1976.10403794. No abstract available. PMID 1246970
- [Background] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Background] Guenther U, Popp J, Koecher L, Muders T, Wrigge H, Ely EW, Putensen C. Validity and reliability of the CAM-ICU Flowsheet to diagnose delirium in surgical ICU patients. J Crit Care. 2010 Mar;25(1):144-51. doi: 10.1016/j.jcrc.2009.08.005. Epub 2009 Oct 13. PMID 19828283
- [Background] McCusker J, Cole MG, Voyer P, Monette J, Champoux N, Ciampi A, Vu M, Belzile E. Six-month outcomes of co-occurring delirium, depression, and dementia in long-term care. J Am Geriatr Soc. 2014 Dec;62(12):2296-302. doi: 10.1111/jgs.13159. Epub 2014 Dec 8. PMID 25482152